CLINICAL TRIAL: NCT05879068
Title: A Phase II Study to Evaluate Efficacy, Safety and Pharmacokinetics of PM8002 Injection in Combination With Paclitaxel Injection as Second Line Treatment for Small Cell Lung Cancer(SCLC)
Brief Title: A Study of PM8002 in Combination With Chemotherapy in Patients With SCLC
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Biotheus Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PM8002-B002C-SCLC-R
Record Dates: First submitted 2023-05-17; First posted 2023-05-30 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: SCLC
Keywords: Second line
MeSH Terms: interventions — Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PM8002+Paclitaxel (Experimental): Subjects will be administered with PM8002 plus Paclitaxel via intravenously (IV) Q3W for 5 cycles, followed by PM8002 until disease progression or intolerable toxicity for a maximum of 2 years.
  Interventions: Drug: PM8002; Drug: Paclitaxel

INTERVENTIONS:
Drug: PM8002 — IV infusion
Drug: Paclitaxel — IV infusion

SUMMARY:
PM8002 is a bispecific antibody targeting PD-L1 and VEGF. This study will evaluate the efficacy and safety of PM8002 in combination with paclitaxel as second line treatment for SCLC.

DETAILED DESCRIPTION:
This is a phase II, single arm study assessing the efficacy and safety of PM8002 in combination with paclitaxel as second line treatment for SCLC who failed first-line platinum-based chemotherapy with or without checkpoint inhibitors therapy

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form before any trial-related processes;
2. Age ≥18 years;
3. Histologically or cytologically confirmed SCLC;
4. Advanced SCLC who failed first-line platinum-based chemotherapy with or without checkpoint inhibitors;
5. Have adequate organ function;
6. The Eastern Cancer Cooperative Group (ECOG) performance score of 0 or 1;
7. Life expectancy of ≥12 weeks;
8. Had at least one measurable tumor lesion according to RECIST v1.1.

Exclusion Criteria:

1. History of severe allergic disease, severe drug allergy or have known allergy to any component of the study drugs;
2. Evidence and history of severe bleeding tendency;
3. History of severe cardiovascular diseases within 6 months;
4. Current presence of severe superior vena cava syndrome and spinal cord compression;
5. Current presence of uncontrolled pleural, pericardial, and peritoneal effusions;
6. History of allogeneic hematopoietic stem cell transplantation or allogeneic organ transplantation;
7. History of alcohol abuse, psychotropic substance abuse or drug abuse;
8. Human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome;
9. Pregnant or lactating women;
10. Other conditions considered unsuitable for this study by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2022-05-27 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | Up to approximately 2 years
  Objective response rate (ORR) is the proportion of subjects with complete response (CR) or partial response (PR), based on RECIST v1.1.
Treatment related adverse events (TRAEs) | Up to 30 days after last treatment
  The incidence and severity of TRAEs graded according to NCI-CTCAE v5.0

SECONDARY OUTCOMES:
Disease control rate (DCR) | Up to approximately 2 years
  DCR is defined as the proportion of subjects with CR, PR, or stable disease(SD) based on RECIST v1.1.
Duration of response (DoR) | Up to approximately 2 years
  DoR is defined as the duration from the first documentation of objective response to the first documented disease progression (based on RECIST v1.1) or death due to any cause, whichever occurs first.
Progression free survival (PFS) | Up to approximately 2 years
  PFS is defined as the time from the start of treatment until the first documentation of disease progression or death due to any cause, whichever occurs first (based on RECIST v1.1).
Overall survival (OS) | Up to approximately 2 years
  OS is the time from the date of first dosing date to death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Cheng, Principal Investigator — Jilin Provincial Tumor Hospital
Locations (11):
- China (11):
  - Peking University Cancer Hospital, Beijing
  - Jilin Provincial Tumor Hospital, Changchun
  - Hunan Cancer Hospital, Changsha
  - Sichuan Provincial People's Hospital, Chengdu
  - Zhejiang Provincial People's Hospital, Hangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - Shandong Cancer Hospital, Jinan
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - Shanghai Pulmonary Hospital, Shanghai
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - Henan Cancer Hospital, Zhengzhou

IPD SHARING:
Plan to Share IPD: Yes
The data will be published or presented for publications (poster, abstract,articles or papers) or any presentations.
Time Frame: After the trial completed.
Access Criteria: NCI is committed to sharing data in accordance with NIH policy.